CLINICAL TRIAL: NCT04116710
Title: A Phase I, First-in-human, Dose-escalation Study to Evaluate the Safety and Immunologic Response After Administration of HS-130 in Combination With HS-110 (Viagenpumatucel-L) in Patients With Solid Tumors Refractory to Standard Care
Brief Title: A Phase 1 Study of HS130 in Combination With Viagenpumatucel-L (HS110) in Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Heat Biologics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS130-001
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Results first posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2022-10

CONDITIONS: Advanced Solid Tumor
Keywords: Cancer; Immunotherapy; Vaccine; Intradermal; gp96; OX40; Combination Therapy; Co-stimulation; Heat Biologics
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1: HS-130 + HS-110 (viagenpumatucel-L) (Experimental): Patients will receive a combination of intradermal HS-130 and HS-110 once every 14 days. The dose levels will be determined by the starting dose and the escalation steps outlined in the protocol.
  Interventions: Biological: HS-110 (viagenpumatucel-L); Biological: HS-130

INTERVENTIONS:
Biological: HS-110 (viagenpumatucel-L) — Vaccine derived from irradiated human lung cancer cells genetically engineered to continually secrete gp96-Ig
Biological: HS-130 — Vaccine derived from irradiated human lung cancer cells expressing the co-stimulatory fusion protein OX40L-Ig

SUMMARY:
This is a phase 1 open-label, single center, dose escalation study to determine a safe and effective maximum tolerated dose of HS-130 in combination with viagenpumatucel-L (HS-110) for adult subjects with advanced solid tumors who are refractory to Standard of Care.

DETAILED DESCRIPTION:
This is an open-label, non-controlled, first-in-human Phase I study of HS-130 and HS-110 in patients with advanced solid tumors refractory to, or ineligible for, Standard of Care.

Seven dose levels will be explored in escalating doses. For each dose level, patients will receive combination HS-130 and HS-110 via intradermal injections once every 14 days. The Dose Limiting Toxicity (DLT) window of observation will include the first 28 days of treatment. In the absence of progressive disease or unacceptable toxicity, patients will continue to receive combination treatment every two weeks until disease progression, death, patient's withdrawal of consent, Investigator decision to discontinue treatment, or intolerable toxicity, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with metastatic or advanced, unresectable solid tumor who have progressed, or recurred following standard-of-care (SOC) therapies or are ineligible for safe and effective SOC therapies and for whom, in the opinion of the Investigator, experimental therapy with HS-130/HS-110 may be beneficial.
2. Patients should have lesions that are safely accessible for biopsy and be willing to provide pre-treatment and on-treatment tissue biopsy. Fine-needle aspiration biopsy is not acceptable. Archival tumor tissue will be accepted in lieu of fresh biopsy at screening if sample was collected within 6-months from Cycle 1 Day 1, and the local pathologist confirms that an adequate amount of tissue/tumor cells exist to allow completion of all testing as outlined in the specimen collection manual.
3. Age ≥ 18 years.
4. Have an acceptable organ function:

   * Albumin ≥ 2.5 g/dL.
   * Total Bilirubin < 3.0 × upper limit of normal (ULN) unless patient has Gilbert's syndrome.
   * Alanine transaminase (ALT) and aspartate transaminase (AST) ≤ 3.0 × ULN or ≤ 5 × ULN in the case of liver metastases.
   * Calculated or measured creatinine clearance > 35 mL/minute per the Cockcroft-Gault formula.
   * Absolute neutrophil count ≥ 1,500/mm3.
   * Hemoglobin ≥ 9 g/dL.
   * Platelet count ≥ 100,000/mm3.
5. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
6. Life expectancy of at least three months.
7. Patients, both females and males, of childbearing/reproductive potential must agree to use adequate contraception while included in the trial and for six months after the last treatment with HS-130 and/or HS-110.
8. Patients must be willing and have the capacity to sign the informed consent form.

Exclusion Criteria:

1. Have clinically significant cardiac disease, including:

   * Onset of unstable angina within 6 months of signing the Informed Consent Form (ICF).
   * Acute myocardial infarction within 6 months of the signing the ICF.
   * Known congestive heart failure (Grade III or IV as classified by the New York Heart Association); and/ or a known decreased cardiac ejection fraction (LVEF) of < 45%.
   * Uncontrolled hypertension defined as systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥ 100 mmHg, despite optimal medical management.
2. Known or clinically suspected leptomeningeal disease. Stable, previously treated metastases in the brain or spinal cord, are allowed as long as these are considered stable (by CT or MRI), and not requiring systemic corticosteroids.
3. History of ≥ grade 3 allergic reactions as well as known or suspected allergy or intolerance to any agent given in the course of this trial, live cell therapies, or live vaccines.
4. History of suspected cytokine release syndrome (CRS).
5. Known immunodeficiency disorders (testing not required).
6. Ongoing or current autoimmune disease. Permanent but stable and manageable immune related adverse events (irAE) from prior therapies are permissible, if prednisone equivalent corticosteroid use does not exceed 10 mg/day.
7. Any other condition requiring concurrent systemic immunosuppressive therapy (other than allowable exceptions which do not exceed 10mg/day of prednisone/corticosteroid use).
8. Major surgery (requiring general anesthesia or inpatient hospitalization) within four weeks before first IMP administration.
9. Any ongoing anticancer therapy including; small molecules, immunotherapy, chemotherapy, monoclonal antibodies or any other experimental drug. Prior therapy must be stopped within four weeks before first infusion in the study, or 5 half-lives, or twice the duration of the biological effect of the investigational product (whichever is shortest). Adjuvant anti-hormonal treatment(s) for previously treated breast cancer or prostate cancer are allowed. Bisphosphonates are allowed, Denosumab and other RANK ligand inhibitors are prohibited.
10. Known current malignancy other than inclusion diagnosis. Prior curable cancer with complete remission for >2 years is allowed.
11. Any other ongoing significant, uncontrolled medical condition as per Investigator discretion.
12. Received a live vaccine within 30 days prior to first dose of study drug.
13. Clinically significant active viral, bacterial or fungal infection requiring:

    1. Intravenous treatment with antimicrobial therapy completed less than two weeks prior to first dose, or
    2. Oral treatment with antimicrobial therapy completed less than one week prior to first dose.

    Prophylactic treatment with antibiotics (e.g. for dental extractions) is allowed.
14. Known positive serology for human immunodeficiency virus (HIV), hepatitis B, or hepatitis C (except in cases of immunity after cured infection). Testing not required.
15. Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the trial or evaluation of the trial result in the opinion of the Investigator.
16. Women who are pregnant or breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-08-12 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel E. Sanborn, MD, Principal Investigator — Providence Cancer Institute
Locations (1):
- Providence Portland Medical Center, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: HS-130 (150 ng- 600 ng) + HS-110 (150 ng - 300 ng) (Viagenpumatucel-L); Cohort 2: HS-130 (600 ng) + HS-110 (600 ng) (Viagenpumatucel-L); Cohort 3: HS-130 (1200 ng) + HS-110 (600 ng) (Viagenpumatucel-L); Cohort 4: HS-130 (1200 ng) + HS-110 (1200 ng) (Viagenpumatucel-L): Patients will receive a combination of intradermal HS-130 and HS-110 once every 14 days. The dose levels will be determined by the starting dose and the escalation steps outlined in the protocol.
  HS-110 (viagenpumatucel-L): Vaccine derived from irradiated human lung cancer cells genetically engineered to continually secrete gp96-Ig
  HS-130: Vaccine derived from irradiated human lung cancer cells expressing the co-stimulatory fusion protein OX40L-Ig
Period: Overall Study
Arm/Group | Cohort 1: HS-130 (150 ng- 600 ng) + HS-110 (150 ng - 300 ng) (Viagenpumatucel-L) | Cohort 2: HS-130 (600 ng) + HS-110 (600 ng) (Viagenpumatucel-L) | Cohort 3: HS-130 (1200 ng) + HS-110 (600 ng) (Viagenpumatucel-L) | Cohort 4: HS-130 (1200 ng) + HS-110 (1200 ng) (Viagenpumatucel-L)
Started | 4 | 6 | 3 | 2
Disease Progression | 4 | 6 | 2 | 2
Completed | 0 | 0 | 0 | 0
Not Completed | 4 | 6 | 3 | 2
Not completed — Death | 4 | 6 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: HS-130 (150 ng- 600 ng) + HS-110 (150 ng - 300 ng) (Viagenpumatucel-L) | Cohort 2: HS-130 (600 ng) + HS-110 (600 ng) (Viagenpumatucel-L) | Cohort 3: HS-130 (1200 ng) + HS-110 (600 ng) (Viagenpumatucel-L) | Cohort 4: HS-130 (1200 ng) + HS-110 (1200 ng) (Viagenpumatucel-L) | Total
Number analyzed (Participants) | 4 | 6 | 3 | 2 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (3.51) | 49.8 (7.52) | 62.3 (7.02) | 69.0 (9.90) | 61.2 (12.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 3 | 0 | 8
  Male | 1 | 4 | 0 | 2 | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 4 | 5 | 3 | 2 | 14
  Race: Unknown | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 4 | 6 | 3 | 2 | 15

OUTCOME MEASURES:

1. Primary Outcome: Dose Limiting Toxicity
Description: Number of Patients with Dose Limiting Toxicity (DLT)
Time Frame: 1 month
Population: The safety population includes all patients who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: HS-130 (150 ng- 600 ng) + HS-110 (150 ng - 300 ng) (Viagenpumatucel-L) | Cohort 2: HS-130 (600 ng) + HS-110 (600 ng) (Viagenpumatucel-L) | Cohort 3: HS-130 (1200 ng) + HS-110 (600 ng) (Viagenpumatucel-L) | Cohort 4: HS-130 (1200 ng) + HS-110 (1200 ng) (Viagenpumatucel-L)
Number analyzed (Participants) | 4 | 6 | 3 | 2
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from Cycle 1 day 1 (first dose) until 30 days after last dose. The study duration was 18 months.
Description: Toxicity was graded per the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v4.03
Arm/Group | Cohort 1: HS-130 (150 ng- 600 ng) + HS-110 (150 ng - 300 ng) (Viagenpumatucel-L) | Cohort 2: HS-130 (600 ng) + HS-110 (600 ng) (Viagenpumatucel-L) | Cohort 3: HS-130 (1200 ng) + HS-110 (600 ng) (Viagenpumatucel-L) | Cohort 4: HS-130 (1200 ng) + HS-110 (1200 ng) (Viagenpumatucel-L)
All-Cause Mortality (participants affected / at risk) | 4/4 | 6/6 | 3/3 | 1/2
Serious Adverse Events (participants affected / at risk) | 0/4 | 1/6 | 1/3 | 1/2
Other Adverse Events (participants affected / at risk) | 4/4 | 6/6 | 3/3 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: HS-130 (150 ng- 600 ng) + HS-110 (150 ng - 300 ng) (Viagenpumatucel-L) (N=4) | Cohort 2: HS-130 (600 ng) + HS-110 (600 ng) (Viagenpumatucel-L) (N=6) | Cohort 3: HS-130 (1200 ng) + HS-110 (600 ng) (Viagenpumatucel-L) (N=3) | Cohort 4: HS-130 (1200 ng) + HS-110 (1200 ng) (Viagenpumatucel-L) (N=2)
Intestinal Ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteremia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Embolic Stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: HS-130 (150 ng- 600 ng) + HS-110 (150 ng - 300 ng) (Viagenpumatucel-L) (N=4) | Cohort 2: HS-130 (600 ng) + HS-110 (600 ng) (Viagenpumatucel-L) (N=6) | Cohort 3: HS-130 (1200 ng) + HS-110 (600 ng) (Viagenpumatucel-L) (N=3) | Cohort 4: HS-130 (1200 ng) + HS-110 (1200 ng) (Viagenpumatucel-L) (N=2)
Fatigue (General disorders) | 3 (3) | 4 (4) | 2 (2) | 1 (1)
Injection Site Pruritus (General disorders) | 2 (2) | 3 (3) | 2 (2) | 1 (1) — general disorders and administration site reactions
Injection Site Erythema (General disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1) — general disorders and administration site reactions
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 4 (4) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/10/NCT04116710/Prot_SAP_000.pdf